CLINICAL TRIAL: NCT06772155
Title: A Comparative Effectiveness Study on Catheter Locking Device Versus Standard Ventriculostomy for Surgical Management of Traumatic Brain Injury Patients With Intracranial Compartment Syndrome
Brief Title: Security and Effectiveness Assessment of Locking Systems in Ventriculostomy for Traumatic Brain Injury
Acronym: SEALS-TBI
Status: Not yet recruiting | Type: Observational
Sponsor: Meditech Foundation (Other)
Responsible Party: Principal Investigator, Andres M. Rubiano, Principal Investigator, Meditech Foundation
Other Study IDs: CEIM-2024-12-101
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Traumatic Brain Injuries; Intracranial Hypertension
Keywords: External Ventricular Drain; Traumatic Brain Injury; Cranial Compartment Syndrome
MeSH Terms: conditions — Brain Injuries, Traumatic; Intracranial Hypertension | interventions — Ventriculostomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Standard Ventriculostomy: Patients are managed with a standard ventriculostomy procedure connected to an external ventricular drain system.
  Interventions: Procedure: Ventriculostomy
- Ventriculostomy + Locking Device: Patients are managed with a ventriculostomy procedure plus a locking system (NTDrain) connected to an external ventricular drain system.
  Interventions: Procedure: Ventriculostomy + Locking Device

INTERVENTIONS:
Procedure: Ventriculostomy — Involves inserting a catheter into the brain's ventricular system to drain cerebrospinal fluid (CSF) and reduce intracranial pressure (ICP). This is a common procedure performed in this type of patient. It can be performed by a frontal approach, using a standard point 10cm from the nasion and 3cm lateral to the midline in the skull. A burr hole is performed and then the catheter is inserted in the frontal horn of the ventricular system. Then the catheter is tunneled subcutaneously and connected to an external ventricular drain collection system that allows also ICP measurement.
  Other Names: Intraventricular Catheter; External Ventricular Drainage
  Groups: Standard Ventriculostomy
Procedure: Ventriculostomy + Locking Device — Involves inserting a catheter into the brain's ventricular system to drain cerebrospinal fluid (CSF) and reduce intracranial pressure (ICP). This is an alternative procedure performed for this type of patient. It can be performed by a frontal approach, using a standard point 10cm from the nasion and 3cm lateral to the midline in the skull. A burr hole is performed and then the catheter is inserted in the frontal horn of the ventricular system. During the insertion, a locking device is attached and secured at the burr hole defect. Then the catheter is tunneled subcutaneously and connected to an external ventricular drain collection system that allows also ICP measurement.
  Other Names: Ventricular Drainage + Locking Device; External Ventricular Catheter + Locking Device
  Groups: Ventriculostomy + Locking Device

SUMMARY:
This study aims to compare the effectiveness and safety of a standard intervention called ventriculostomy for managing increased intracranial pressure (ICP) in patients with severe traumatic brain injury (TBI). Elevated ICP is a critical condition that can result in brain damage or death if not treated promptly. The intervention will be performed in a traditional standard way or with an additional device called a catheter locking system. The first approach, standard ventriculostomy, involves placing a catheter into the brain's ventricular system to drain cerebrospinal fluid (CSF), thereby reducing ICP. The second approach incorporates the same catheter plus a catheter-locking device designed to secure the catheter in place, potentially reducing complications such as catheter displacement and the need for additional surgeries. Participants in this study will undergo either standard ventriculostomy or ventriculostomy with the locking device. Their progress will be observed during their hospital stay until the catheter is taken out (regularly on days 5th to 7th after the initial surgery) and assessed over one year through structured telephone follow-ups. The main outcomes include functional recovery, as measured by the Glasgow Outcome Scale Extended (GOSE), and the rate of complications such as operative site infections, catheter displacement, and/or reinterventions. By comparing these two methods, the study seeks to determine whether the locking device improves outcomes for TBI patients while maintaining or enhancing the safety and reliability of the procedure.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) patients often exhibit an increase in their intracranial volume due to blood collection or brain tissue edema. When the volume of any intracranial compartment exceeds a critical threshold, the compensatory mechanisms become overwhelmed, compromising intracranial compliance and blood supply, which leads to intracranial compartment syndrome (ICCS) and further exacerbates brain damage through secondary injury. When less invasive measures to counteract ICCS prove insufficient, ventriculostomy connected to an external ventricular drainage system is a treatment option, where positioning an intraventricular catheter by the frontal horn of the lateral ventricles is the preferred technique. Although its effectiveness has been demonstrated, ventriculostomy is also associated with a high incidence of complications. Locking devices for decreasing the movement of the catheter have been proposed as an alternative that leverages the benefits of ventriculostomy while reducing the associated adverse effects.

This study will compare the functional outcomes and complications linked to ventriculostomy and the use of locking devices for the ventricular catheter. Standard Ventriculostomy: Involves inserting a catheter into the brain's ventricular system to drain cerebrospinal fluid (CSF) and reduce intracranial pressure (ICP). This is a common procedure performed in patients with traumatic brain injury who request invasive ICP monitoring and/or CSF drainage.

The Ventriculostomy with a Locking Device is the same procedure, but it will be performed with an additional approved device, a locking system that secures the catheter in place, reducing the risk of displacement and associated complications. The system requires internal approval by regulatory entities in each one of the participant countries. Most of them already have approval and the others are in an internal approval process. Countries cannot start collecting data until they have the internal government approval for the device distribution by internal medical suppliers.

ELIGIBILITY:
Inclusion Criteria:

1. TBI patients arriving at the emergency room in the first 24 hours following trauma.
2. Abnormal Computed Tomography (CT), with a primary injury including any epidural, intracerebral, or subdural collection with a midline shift >3 mm and any basal cistern compression with at least 2 abnormal findings in the initial evaluation at the emergency room (including optic nerve ultrasound > 6mm on the same side of the CT´s primary injury and/or an abnormal pupillometry with a reduced Maximum Contraction Velocity (MCV) in the pupil of the same side of the CT´s primary injury, or/and a Trans-Cranial Doppler (TCD) with Pulsatility Index (PI) > 1.3 and/or Medium Cerebral Artery - Diastolic Velocity (MCA-DV) < 20cm/seg on the same side of the CT´s primary injury or/and an Intracranial Pressure Wave Form (ICPWF)2 > ICPWF1 waveform pattern on the same side of the CT´s primary injury).
3. Age 18 to 70 years old.
4. Patients with or without polytrauma with survival expectancy >24 hours.
5. Ventriculostomy surgical procedures less than 24 hours after the trauma.

Exclusion Criteria:

1. TBI patients arriving at the emergency room after 24 hours following trauma.
2. Normal CT scan at the emergency room.
3. Abnormal CT scan at the emergency room with any primary injury and midline shift less than 3mm or without basal cistern compression and with normal values in at least two different modalities of assessing ICCS (pupillometry, optic nerve sheath ultrasound, transcranial Doppler, and/or non-invasive ICP waveform analyzer).
4. Age less than 18 or more than 70 years old.
5. Polytrauma or massive brain injury with survival expectancy < 24 hours.
6. Ventriculostomy surgical procedures performed > 24 hours after the trauma.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients arriving at any of the recruitment centers (tertiary hospitals or level
  1 hospitals / specialized hospitals) in any of the involved countries (Bolivia, Brazil, Cambodia, Cameroon, Chile, Colombia, Dominican Republic, Ecuador, Egypt, Guatemala, Italy, Nigeria, Paraguay, Peru, Philippines, Rwanda, Serbia, Tanzania, Thailand, Venezuela).
Sampling Method: Non-Probability Sample
Enrollment: 292 (Estimated)
Dates: Start 2025-07-05 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
GOSE | 12 months
  Extended Glasgow Outcome Scale, evaluated from 1 to 8 points without dichotomization, with 1 being the worst outcome and 8 being the best outcome.

SECONDARY OUTCOMES:
Ventriculostomy Related Complications | 15 days.
  Complications of the post-operative period related to displacements, infection, CSF disturbances, obstruction, and other technical (ICP misreadings) and medical problems associated with the intraventricular catheter.

CONTACTS AND LOCATIONS:
Overall Officials: Andres M Rubiano, MD, Principal Investigator — Meditech Foundation; Luigi V Berra, MD, Principal Investigator — La Sapienza University

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analyzed during the current study will be available upon request to the key personnel of the sponsor institution. Individual participant data (IPD) will be stored in a private repository and made available upon request. Once requested, the unprocessed data collected on the RedCap platform will be shared as soon as possible. The shared data will be anonymous, as the only identifier will be the ID assigned to patients participating in the study. No additional consents are required for sharing IPD, as this possibility is included in the informed consent.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From June 2025 to June 2027
Access Criteria: The datasets generated during and/or analyzed during the current study will be available upon request to the key personnel of the sponsor institution (see contact information). Individual participant data (IPD) will be stored in a private repository and made available upon request. Once requested, the unprocessed data collected on the RedCap platform will be shared as soon as possible. The shared data will be anonymous, as the only identifier will be the ID assigned to patients participating in the study. No additional consents are required for sharing IPD, as this possibility is included in the informed consent.
URL: http://www.seals-tbi-study.com

REFERENCES:
- [Background] Stuart MJ, Antony J, Withers TK, Ng W. Systematic review and meta-analysis of external ventricular drain placement accuracy and narrative review of guidance devices. J Clin Neurosci. 2021 Dec;94:140-151. doi: 10.1016/j.jocn.2021.10.014. Epub 2021 Oct 26. PMID 34863429
- [Background] Brotis AG, Karvouniaris M, Tzerefos C, Gatos C, Fountas KN. Guidelines on the use of external ventricular drain and its associated complications: do we "AGREE II"? Br J Neurosurg. 2021 Dec;35(6):689-695. doi: 10.1080/02688697.2021.1958153. Epub 2021 Aug 9. PMID 34365868
- [Background] Lele AV, Hoefnagel AL, Schloemerkemper N, Wyler DA, Chaikittisilpa N, Vavilala MS, Naik BI, Williams JH, Venkat Raghavan L, Koerner IP; Representing SNACC Task Force for Developing Guidelines for Perioperative Management of External Ventricular and Lumbar Drains. Perioperative Management of Adult Patients With External Ventricular and Lumbar Drains: Guidelines From the Society for Neuroscience in Anesthesiology and Critical Care. J Neurosurg Anesthesiol. 2017 Jul;29(3):191-210. doi: 10.1097/ANA.0000000000000407. PMID 28169966
- [Background] Fried HI, Nathan BR, Rowe AS, Zabramski JM, Andaluz N, Bhimraj A, Guanci MM, Seder DB, Singh JM. The Insertion and Management of External Ventricular Drains: An Evidence-Based Consensus Statement : A Statement for Healthcare Professionals from the Neurocritical Care Society. Neurocrit Care. 2016 Feb;24(1):61-81. doi: 10.1007/s12028-015-0224-8. PMID 26738503
- [Background] Godoy DA, Brasil S, Rubiano AM. Further support for the intracranial compartmental syndrome concept. Crit Care. 2024 Sep 18;28(1):311. doi: 10.1186/s13054-024-04974-4. No abstract available. PMID 39294706
- [Background] Martinez-Palacios K, Vasquez-Garcia S, Fariyike OA, Robba C, Rubiano AM; noninvasive intracranial pressure monitoring international consensus group. Quantitative Pupillometry for Intracranial Pressure (ICP) Monitoring in Traumatic Brain Injury: A Scoping Review. Neurocrit Care. 2024 Aug;41(1):255-271. doi: 10.1007/s12028-023-01927-7. Epub 2024 Feb 13. PMID 38351298
- [Background] Martinez-Palacios K, Vasquez-Garcia S, Fariyike OA, Robba C, Rubiano AM; noninvasive ICP monitoring international consensus group. Using Optic Nerve Sheath Diameter for Intracranial Pressure (ICP) Monitoring in Traumatic Brain Injury: A Scoping Review. Neurocrit Care. 2024 Jun;40(3):1193-1212. doi: 10.1007/s12028-023-01884-1. Epub 2023 Dec 19. PMID 38114797
- [Background] Martinez-Palacios K, Vasquez-Garcia S, Fariyike OA, Robba C, Rubiano AM. Non-Invasive Methods for Intracranial Pressure Monitoring in Traumatic Brain Injury Using Transcranial Doppler: A Scoping Review. J Neurotrauma. 2024 Jun;41(11-12):1282-1298. doi: 10.1089/neu.2023.0001. Epub 2024 Apr 11. PMID 37861291
- [Background] Godoy DA, Brasil S, Iaccarino C, Paiva W, Rubiano AM. The intracranial compartmental syndrome: a proposed model for acute brain injury monitoring and management. Crit Care. 2023 Apr 10;27(1):137. doi: 10.1186/s13054-023-04427-4. PMID 37038236
- [Background] Rubiano AM, Figaji A, Hawryluk GW. Intracranial pressure management: moving beyond guidelines. Curr Opin Crit Care. 2022 Apr 1;28(2):101-110. doi: 10.1097/MCC.0000000000000920. PMID 35058406
- [Background] Rubiano AM, Griswold DP, Jibaja M, Rabinstein AA, Godoy DA. Management of severe traumatic brain injury in regions with limited resources. Brain Inj. 2021 Sep 19;35(11):1317-1325. doi: 10.1080/02699052.2021.1972149. Epub 2021 Sep 7. PMID 34493135
- [Background] Hawryluk GWJ, Aguilera S, Buki A, Bulger E, Citerio G, Cooper DJ, Arrastia RD, Diringer M, Figaji A, Gao G, Geocadin R, Ghajar J, Harris O, Hoffer A, Hutchinson P, Joseph M, Kitagawa R, Manley G, Mayer S, Menon DK, Meyfroidt G, Michael DB, Oddo M, Okonkwo D, Patel M, Robertson C, Rosenfeld JV, Rubiano AM, Sahuquillo J, Servadei F, Shutter L, Stein D, Stocchetti N, Taccone FS, Timmons S, Tsai E, Ullman JS, Vespa P, Videtta W, Wright DW, Zammit C, Chesnut RM. A management algorithm for patients with intracranial pressure monitoring: the Seattle International Severe Traumatic Brain Injury Consensus Conference (SIBICC). Intensive Care Med. 2019 Dec;45(12):1783-1794. doi: 10.1007/s00134-019-05805-9. Epub 2019 Oct 28. PMID 31659383
- [Background] Chau CYC, Craven CL, Rubiano AM, Adams H, Tulu S, Czosnyka M, Servadei F, Ercole A, Hutchinson PJ, Kolias AG. The Evolution of the Role of External Ventricular Drainage in Traumatic Brain Injury. J Clin Med. 2019 Sep 10;8(9):1422. doi: 10.3390/jcm8091422. PMID 31509945
- [Background] Carney N, Totten AM, O'Reilly C, Ullman JS, Hawryluk GW, Bell MJ, Bratton SL, Chesnut R, Harris OA, Kissoon N, Rubiano AM, Shutter L, Tasker RC, Vavilala MS, Wilberger J, Wright DW, Ghajar J. Guidelines for the Management of Severe Traumatic Brain Injury, Fourth Edition. Neurosurgery. 2017 Jan 1;80(1):6-15. doi: 10.1227/NEU.0000000000001432. PMID 27654000